CLINICAL TRIAL: NCT05703321
Title: The Relationship of Preoperative Fasting With Tricuspid Annular Plane Systolic Movement in Female Patients
Acronym: FASTİNGTAPSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aydin Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, Anesthesiologist, Aydin Maternity and Child Health Hospital
Other Study IDs: 2022/185
Record Dates: First submitted 2023-01-13; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: TAPSE
Keywords: Preoperative Fasting; volume; Tricuspid Annular Plane Systolic Movement; right ventricle function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: preoperative fasting — Fasting for 6 hours is required for the patients regarding the preparation of the operation and preparation for anesthesia

SUMMARY:
Background Fasting for 6 hours is required for the patients regarding the preparation of the operation and preparation for anesthesia. It is already known that this fasting period affects volume. Although Tricuspid Annular Plane Systolic Movement (TAPSE) is an echocardiographic parameter showing Right Ventricular (RV) systolic function, its relationship with volume is discussed in recent years. In the present study, the relationship between TAPSE and volume, and whether there is a change in preoperative fasting and right ventricular functions will be evaluated.

Methods The study was started between 21.11.2022 and 21.05.2023 in Aydın Maternity and Child Hospital after approval was received from the Non-Invasive Clinical Research Ethics Committee. A total of 21 patients were planned to be included in this prospective observational study. Transthoracic echocardiography will be performed in patients aged 18-65 years who will undergo elective procedures under anesthesia, and in full patients the day before surgery. Those who are pregnant, patients with known or prospective severe valvular disease, severe pulmonary hypertension, acute myocardial infarction, dilated and hypertrophic cardiomyopathy, and non-sinus rhythm will be excluded from the study. Transthoracic echocardiography will be performed on the patients, and the relationship between TAPSE and volume and whether there is a change in preoperative fasting and right ventricular functions will be evaluated.

DETAILED DESCRIPTION:
It is already known that right ventricular systolic dysfunction has prognostic value in various pathological conditions. Evaluating RV function with echocardiography is difficult because of the complex geometry of the RV. Although RV function was evaluated only visually for many years, guidelines have been published by the American Society of Echocardiography as a result of studies conducted in recent years. In this respect, abnormal RV function must be suspected in case of one of the following criteria S'<10 cm/s, TAPSE <16 mm, RVFAC <35%, or R-MPI (tissue Doppler) > 0.55. Combining multiple measures of RV function can more reliably distinguish normal from abnormal function. TAPSE is a parameter that can be easily measured for apex-basal shortening and gives specific information about the global RV function. When compared to other measures of RV function, it is less dependent on optimal image quality and easier to measure. Low TAPSE is not very common but has been measured in some individuals without heart disease because of measurement errors, diagnostic misclassification, and extremes of the normal spectrum. It was shown in the study conducted by Gullupınar et al. that TAPSE decreased significantly after blood donation in people who had donated blood. Also, studies are trying to determine a relationship between central venous pressure, which is a volume indicator, and TAPSE. There is also a study that reported a relationship between cardiac MRI and CT and the right ventricle.

The purpose of the present study is to try to correlate the volume change of TAPSE because of preoperative hunger and to determine whether there is a change in preoperative fasting and right ventricular functions.

Purpose: To show whether there is a relationship between volume and TAPSE. To determine the relationship of TAPSE with preload and its usability for this purpose, and whether there is a change in preoperative fasting and right ventricular functions.

Hypothesis: TAPSE value is related to volume.

Material Method The study will start between 21.11.2022 and 21.05.2023 in Aydın Maternity and Child Hospital, after the approval of the Non-Invasive Clinical Research Ethics Committee. Measurements will be made and recorded with Transthoracic Echocardiography (TTE) one day before the surgery, and TTE again if the preoperative fasting times on the day of the operation are appropriate in patients aged between 18-65 years who will undergo elective procedures under anesthesia. TTE will be made by the principal investigator Ferdi GULASTI. The demographic characteristics of the patients, preoperative blood values, heart rate during TTE, oxygen saturation (SaO2), Systolic Arterial Pressure (SAP), Diastolic Arterial Pressure (DAP), and Mean Arterial Pressure (MAP) will be recorded. The data will be compared statistically after the data collection process for the study is completed.

Echocardiography TTE will be performed on all patients in the left lateral decubitus position with the Echocardiography Device by the same observer. The values of all parameters will be recorded by taking the mean values of three cardiac cycle measurements. The measurement methods will be performed in line with the Guidelines of the American Society of Echocardiography. M-Mode, 2D (2D) images, color, pulse, and Continuous Wave Doppler and Tissue Doppler measurements will be taken from all participants in line with standard echocardiographic application methods. LV Ejection Fraction (EF) measurements will be evaluated in the parasternal long-axis view.

FACs, S' rates, TAPSE scores, and TDI-derived Myocardial Performance Indices (MPI) will be measured to assess Right Ventricular (RV) systolic functions. Tricuspid E and A wave velocity, E/A ratio, and E' velocity will be measured to assess the diastolic function of the RV. TAPSE will be calculated by placing an M-mode cursor across the Tricuspid Ring and measuring the amount of longitudinal movement in peak systole. Annular peak systolic velocity (S), early (E'), and late (A') peak annular diastolic velocities, Ejection Time (ET), IVRT, and Isovolumetric Contraction Time (IVCT) will be measured from the TDI images. TDI-induced MPI will be calculated as the sum of IVCT and IVRT divided by ET (MPI = (IVRT + IVCT) / ET) as a global estimate of both the systolic and diastolic functions of the RV.

The patients will be visualized in the supine position and through the subxiphoid window of the Inferior Vena Cava (IVC). The cursor will be placed 1 cm distal to the hepatic vein IVC entry point and the IVC diameter will be monitored for 30 seconds in M-Mode. The measurement will be made from the region where the diameter of the inferior vena cava is in inspiration (IVCins) and expiration (IVCexp) while the patient is breathing normally. The Inferior Vena Cava Depression Rate (IVC-CI) will be calculated by using the formula IVC-CI = (IVCexp - IVCins)/IVCexp.

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1-2
2. Being between the ages of 18-65
3. Having no peroperative hydration
4. Preoperative sedative not given
5. No known heart disease

Exclusion Criteria:

1. Being pregnant
2. Post cardiac surgery
3. Severe pulmonary hypertension
4. Severe valve disease
5. Hypertrophic or dilated cardiomyopathy
6. Presence of acute myocardial infarction
7. Non-sinus rhythm

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — because , our hospital is maternity hospital.
Study Population: who will undergo elective procedures under anesthesia
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-05-21 (Estimated); Study Completion 2023-05-21 (Estimated)

PRIMARY OUTCOMES:
TAPSE volume | 6 month
  TAPSE, which is the right ventricular systolic function value, decreases after fasting, which is desired before the surgery

SECONDARY OUTCOMES:
fasting RV function | 6 month
  fasting is related to RV function

CONTACTS AND LOCATIONS:
Locations (1):
- Aydin Maternity and Child Health Hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
study protocol and statistical analysis available to other researchers